CLINICAL TRIAL: NCT02769702
Title: Prospective Open Label Study of Acthar SQ Gel Injection in Patients With Active Anterior Uveitis Who Are Not Well Controlled With, or Intolerant of, Topical or Systemic Corticosteroids
Brief Title: Open Label Study of Acthar SQ Gel Injection in Patients With Active Anterior Uveitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acthar Uveitis Study
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Uveitis
Keywords: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Acthar 80 IU SC twice w eek
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Acthar 80 IU SC twice a week
  Other Names: Acthar Gel

SUMMARY:
Uveitis is an acute or chronic inflammatory condition of unknown etiology. Although uveitis often responds adequately to topical corticosteroids, there are many patients for which this treatment is either inadequate or not tolerated. A patient with inadequate response to treatment would manifest uveitis activity by slit lamp examination determination of anterior chamber cellularity. Lack of tolerance of therapy commonly manifests as ocular hypertension (greater than 21 mmHg measured by tonometry)complicating chronic topical corticosteroid administration, leading to glaucoma and permanent visual loss. Moreover, systemic corticosteroids may be required at a dose unsafe for chronic administration. In these situations, an immunosuppressive medication is often added as a "steroid-sparing" agent. If and when there is clinical response to the added immunosuppressive, the oral and/or topical corticosteroid dose can be reduced or eliminated to avoid toxicity.

There are several reasons for believing that Acthar might be beneficial in the treatment of uveitis patients. In addition to increasing adrenal production or cortisol, Acthar has another important mechanisms of action mediated by its binding of melanocortin receptors. Melanocortin down-regulates activity of B and T lymphocytes, monocytes and macrophages. In animal studies, melanocortin peptides down-regulate T helper cells, up-regulate T Regulatory cells, and decrease B lymphocyte production of B Lymphocyte Stimulator. In macrophages, there is down-regulation of IL-1, IL-2, INF gamma, TNF alpha, nitric oxide and adhesion molecules. In other cells, in addition to IL-10 upregulation (monocytes), there is down-regulation of VACM and ECAM (endothelial cells), prostaglandins (fibroblasts) and MCP-1 and RANTES (renal tubules).CNS mediation of systemic inflammation may also be down-regulated by melanocortin receptor binding by Acthar.

DETAILED DESCRIPTION:
Patients eligible for the study will be identified by the investigators and given a copy of the consent form to read. Patients interested in enrolling will be screened and if eligible will be enrolled in the study. The screening visit and the baseline visit may occur on the same day. Patients enrolling will be instructed in self-administering Acthar 80 IU twice a week. Patients will keep an injection log which will be inspected at each visit (4, 8, and 12 weeks). Ophthalmology data will be collected at each visit and recorded on the case report form by the ophthalmology technician working with the sub-investigator at the time of each visit. Patients will come to the Center for Clinical Studies each visit for blood draw, blood pressure recording, and recording of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Active anterior uveitis requiring oral and/or topical corticosteroid therapy

Exclusion Criteria:

* Uncontrolled diabetes
* Uncontrolled glaucoma
* HIV infection or other infection for which corticosteroid therapy contraindicated
* Contraindication to ACTHAR
* Scleroderma
* Osteoporosis
* Ocular herpes simplex
* Systemic fungal infection
* Recent surgery
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Brasington, MD, Principal Investigator — Washington U Rheumatology
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acthar 80 IU: Acthar 80 IU SC twice week
Period: Overall Study
Arm/Group | Acthar 80 IU
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acthar 80 IU
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eye With Uveitis of Anterior Chamber Cellularity Graded From 0-4 on a Likert Scale Determined by Slit Lamp Examination
Description: standard assessment of uveitis activity. Scores were assessed using a Likert scale using 0 to 4, higher score reflects more cellularity.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acthar 80 IU
Number analyzed (Participants) | 2
units on a scale
  Baseline | 0.5 (0.70)
  12 Weeks | 1.25 (1.06)

2. Secondary Outcome: Change in Baseline in Eye With Uveitis of Anterior Chamber Protein Graded 0-4 on a Likert Scale Determined by Slit Lamp Evaluation
Description: standard assessment of uveitis activity. Scores were assessed using a Likert scale using 0 to 4, higher score reflects more protein.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acthar 80 IU
Number analyzed (Participants) | 2
units on a scale
  Baseline | NA (NA) — Score could not be determined for 1 of the 2 participants.
  12 Weeks | 1.0 (1.41)

ADVERSE EVENTS:
Arm/Group | Acthar 80 IU
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
This study was prematurely terminated, only 2 participants enrolled. Although results are reported they should be interpreted with caution due to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No